CLINICAL TRIAL: NCT01316562
Title: Valeur prédictive d'Une évaluation Cognitive standardisée en Centre d'Examens de Santé Pour le Diagnostic de la Maladie d'Alzheimer ou Des Maladies apparentées en Population générale Chez Les Plus de 65 Ans Avec Plainte mnésique
Brief Title: Predictive Value of Cognitive Tests Performed for the Diagnosis of Alzheimer's Disease and Related Disorders
Acronym: EVATEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Fantino Bruno, Centre d'Examen de Santé de Baraban
Other Study IDs: 2009-025B
Record Dates: First submitted 2011-03-11; First posted 2011-03-16 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Alzheimer's Disease; Impaired Cognition; Memory Disorders
MeSH Terms: conditions — Alzheimer Disease; Cognition Disorders; Memory Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Healthy controls
- Group 2: Patients with an Alzheimer's disease or related disorders

SUMMARY:
The purpose of this study is to determine the predictive value of standardized cognitive tests performed in health examination centres for the diagnosis of Alzheimer's disease and related disorders among adults aged 65 years and older with a subjective memory complaint.

DETAILED DESCRIPTION:
The main objective of this study is to determine the predictive value of standardized cognitive tests performed in health examination centres for the diagnosis of Alzheimer's disease and related disorders among adults aged 65 years and older with a subjective memory complaint.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Community-dwellers
* Volunteers receiving a free medical examination in Health examination centre
* Subjective memory complaint

Exclusion Criteria:

* Known dementia
* Sensory deficit compromising the cognitive evaluation
* Poor workmanship of the written or oral French language

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All subjects with memory complaint recruited during a free medical examination in Health examination centres of Lyon, Saint-Etienne and Angers, France
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Score of episodic memory and executive psychometric tests | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Fantino, Professor, Principal Investigator — CES de Baraban, Lyon
Locations (1):
- CES Baraban, Lyon, France

REFERENCES:
- [Derived] Vannier-Nitenberg C, Dauphinot V, Bongue B, Sass C, Bathsavanis A, Rouch I, Deville N, Beauchet O, Krolak-Salmon P, Fantino B. Performance of cognitive tests, individually and combined, for the detection of cognitive disorders amongst community-dwelling elderly people with memory complaints: the EVATEM study. Eur J Neurol. 2016 Mar;23(3):554-61. doi: 10.1111/ene.12888. Epub 2015 Oct 30. PMID 26518736
- [Derived] Vannier-Nitenberg C, Dauphinot V, Bongue B, Sass C, Rouch I, Beauchet O, Krolak-Salmon P, Fantino B. Early detection of memory impairment in people over 65 years old consulting at Health Examination Centers for the French health insurance: the EVATEM protocol. BMC Geriatr. 2013 Jun 6;13:55. doi: 10.1186/1471-2318-13-55. PMID 23742705